Version 4 Date: 11<sup>th</sup> June 2018 IRAS ID: 230391



## **Informed Consent**

Study Title: An investigation into the feasibility of incorporating an exercise rehabilitation programme for people with intermittent claudication into an already established Cardiac Rehabilitation service

The University of Salford attaches high priority to the ethical conduct of research. We therefore ask you to consider the following points before signing this form. **Your signature confirms you are happy to participate in the study**.

I, the undersigned, confirm that (please initial each box as appropriate):

| 1. | I have read and understood the information about the project, as provided in the Patient Information Sheet dated 11 <sup>th</sup> June 2018 |
|---|---|
| 2. | I have been given the opportunity to ask questions about the project and my participation |
| 3. | I understand I can withdraw at any time without giving reasons and that I will not be penalised for withdrawing nor will I be questioned on why I have withdrawn. I also understand that if I withdraw after the group interview stage, the data I have given up to that point will remain part of the study |
| 4. | The procedures regarding confidentiality have been clearly explained (e.g. use of names, pseudonyms, anonymisation of data, etc.) to me |
| 5. | If applicable, separate terms of consent for interviews, audio, video or other forms of data collection have been explained and provided to me |
| 6. | I agree for my general practitioner (GP) to be informed about my participation in this study |
| 7. | I agree to keep what is discussed in the group interviews confidential |
| 8. | I understand that other researchers will have access to this data only if they agree to preserve the confidentiality of the data and if they agree to the terms I have specified in this form |
| 9. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from University of Salford, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. |
| 10. | The use of the data in research, publications, sharing and archiving has been explained to me, and that only anonymised quotes will be included in publications |

| Participant: | | |
|---------------------|---------------|----------|
| Name of Participant | Signature | <br>Date |
| Researcher: | | |
| Name of Researcher | <br>Signature | <br> |